CLINICAL TRIAL: NCT03516331
Title: A Phase 1, Open Label, Drug-Drug Interaction Study of FDL169 and FDL176 in Healthy Subjects
Brief Title: A Drug-Drug Interaction Study of FDL169 and FDL176 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Flatley Discovery Lab LLC (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FDL169-2017-07
Record Dates: First submitted 2018-04-24; First posted 2018-05-04 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-11

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1:FDL176 & FDL169 coadministration (Experimental): To receive a single dose of FDL176 on Day 1, followed up FDL169 TID starting Day 8; and another single dose of FDL176 on Day 22.
  Interventions: Drug: FDL176 & FDL169 coadministration
- Part 2:FDL176 & FDL169 coadministration (Experimental): To receive FDL176 QD starting Day 1, and FDL169 TID starting Day 8
  Interventions: Drug: FDL176 & FDL169 coadministration

INTERVENTIONS:
Drug: FDL176 & FDL169 coadministration — CFTR corrector and potentiator

SUMMARY:
This is an 2-part study. Part 1 will assess the safety, tolerability and pharmacokinetics of single doses of FDL176 with and without co-administration of FDL169. Part 2 will assess the safety, tolerability and pharmacokinetics of repeated doses of FDL176 with and without co-administration of FDL169 .

DETAILED DESCRIPTION:
This is an open-label, non-randomised, single-sequence 2-part study. Enrolment into Part 2 of the study will begin after Part 1 is complete, and a review of safety and pharmacokinetic data has been completed.Part 1 will assess the safety, tolerability and pharmacokinetics of single doses of FDL176 with and without co-administration of FDL169. Part 2 will assess the safety, tolerability and pharmacokinetics of repeated doses of FDL176 once daily (QD) with and without co-administration of FDL169.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or non-pregnant, non-lactating healthy females.
* Body mass index of 18.0 to 32.0 kg/m2 or, if outside the range, considered not clinically significant by the investigator.
* Must agree to follow the study's contraception requirement

Exclusion Criteria:

* Prior or ongoing medical condition, medical history, physical findings, ECG findings or laboratory abnormality that, in the Investigator's (or delegate's) opinion, could adversely affect the safety of the subject or would place the subject at increased risk.
* History of long QT syndrome and/or QT corrected according to Fridericia's formula (QTcF) interval (>450 msec) or QTcF >450 msec at Screening or Day -1.
* Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hayfever is allowed unless it is active.
* Use of any prescription drugs within 14 days or 5 half-lives (whichever is longer) before the first dose of IMP, unless in the opinion of the Investigator (or delegate) .
* Use of any non-prescription drugs, including vitamins, herbal and dietary supplements within 14 days or 5 half-lives (whichever is longer) before the first dose of IMP.
* Use of any prescription and non-prescription medications that are strong inhibitors or moderate inducers of cytochrome P450 3A, within 28 days before the first dose of IMP.
* Participation in another clinical trial involving receipt of an IMP within the past 90 days.
* Prior exposure to FDL169 or FDL176
* Alkaline phosphatase, aspartate aminotransferase and/or alanine aminotransferase >1.5 x upper limit of normal (ULN) at screening.
* Serum creatinine or total bilirubin >1.5 x ULN (isolated bilirubin >1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin is <35%).
* Abnormal renal function at screening, defined as estimated glomerular filtration rate <60 mL/min using the Modification of Diet in Renal Disease (MDRD) equation.
* History of human immunodeficiency virus (HIV) or positive HIV, hepatitis B or hepatitis C results at screening.
* Positive urinary drugs of abuse screen at Screening or Day -1, or positive alcohol breath test at Screening or Day -1. Consumption of alcohol within 24 h prior to admission.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2018-08-22 (Actual); Study Completion 2018-08-22 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters, Cmax | 72 days
  The pharmacokinetic parameters of FDL176 when co-administered with FDL169, compared to the pharmacokinetics of FDL176 alone; maximal plasma concentration (Cmax)

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 72 days
  Safety and tolerability of FDL176 when co-administered with FDL169, compared to FDL176 alone. as determined by the incidence of adverse events (Aes) and serious adverse events (SAE)s.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Ordonez, MD, Study Chair — Flatley Discovery Lab
Locations (1):
- Quotient Sciences, Nottingham, Ruddington, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided